CLINICAL TRIAL: NCT05373823
Title: A Digital Intervention to Improve Skin Self-examination Among Melanoma Survivors
Brief Title: MySmartSkin Online Skin Self-exam Intervention for Melanoma Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sharon Manne, PhD, Associate Director for Cancer Prevention, Control and Population Science, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: CINJ132202; R01CA264548 (NIH)
Record Dates: First submitted 2022-04-28; First posted 2022-05-13 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Melanoma
Keywords: Self-Examination
MeSH Terms: conditions — Melanoma; Self-Examination

STUDY DESIGN:
Intervention Model Description: Type one hybrid effectiveness-implementation study consisting of three aims. Aim 1 (Months 1-15) focuses on MSS enhancement using stakeholder collaboration. Aim 2 (Months 16-60) involves the longitudinal RCT comparing behavioral outcomes and effectiveness of enhanced MSS versus an educational webpage on SSE as well as new recurrences/melanomas. Aim 3 (Months 16-60) is a mixed-methods study with multi-level stakeholders to assess implementation outcomes and identify contextual factors to facilitate scale-up for future dissemination and implementation. The figure below illustrates the integration of the PHM and implementation science frameworks with the study's aims.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhance MSS using multi-level stakeholder collaboration (Mo.1-15) (Experimental): Enhancements of MSS to increase intervention effects - theory - based strategies (PHM), (BCT)
  Interventions: Other: MySmartSkin enhancement
- Involves the longitudinal RCT comparing behavioral outcomes and effectiveness (Mo.16 -60) (Experimental): RCT of enhanced MSS testing effectiveness (thorough SSE, sun protection behavior Involves the longitudinal RCT comparing behavioral outcomes and effectiveness of enhanced MSS versus an educational webpage on SSE as well as new recurrences/melanomas
  Interventions: Other: Educational webpage on Skin Self-Examination
- Aim 3: Assess implementation outcomes, identify factors relevant for future scale-up (Mo.17-60) (Active Comparator): Assessment of implementation outcomes and key contextual factors from the perspective of multi - level stakeholders
  Interventions: Other: Assess implementation outcomes

INTERVENTIONS:
Other: MySmartSkin enhancement — Focuses on MySmartSkin web application/intervention including enhancements using stakeholder collaboration and input
  Arms: Enhance MSS using multi-level stakeholder collaboration (Mo.1-15)
Other: Educational webpage on Skin Self-Examination — Longitudinal RCT comparing behavioral outcomes and effectiveness of enhanced MSS versus an educational webpage on SSE as well as new recurrences/melanomas
  Arms: Involves the longitudinal RCT comparing behavioral outcomes and effectiveness (Mo.16 -60)
Other: Assess implementation outcomes — A mixed-methods study with multi-level stakeholders to assess implementation outcomes and identify contextual factors to facilitate scale-up for future dissemination and implementation.
  Arms: Aim 3: Assess implementation outcomes, identify factors relevant for future scale-up (Mo.17-60)

SUMMARY:
This project, mySmartSkin (MSS), includes an innovative Type 1 hybrid effectiveness-implementation trial designed to enhance the effects of MSS and simultaneously assess key implementation outcomes (e.g., cost, adoption) as well as contextual factors important for scale-up in community and health care settings where melanoma survivors receive follow-up care. A type 1 hybrid effectiveness-implementation design allows us to engage multilevel stakeholders throughout this process, evaluate the effectiveness of the enhanced MSS, and identify critical factors for wide-scale implementation. Aim 1 will focus on enhancing the previous version of MSS by collaborating with multi-level stakeholders in qualitative interviews and usability testing. Aim 2 will evaluate the effects of enhanced MSS on thorough skin-self examinations (SSE) in a randomized-control trial (RCT) and examine its impact on the diagnosis of new/recurrent melanomas. Aim 3 will focus on assessing selected implementation outcomes and identify factors relevant to future scale-up for widespread dissemination and implementation.

DETAILED DESCRIPTION:
This is a type one hybrid effectiveness-implementation study consisting of three aims. Aim one (Months 1-15) focuses on MSS enhancement using stakeholder collaboration. Aim two (Months 16-60) involves the longitudinal randomized control trial (RCT) comparing behavioral outcomes and effectiveness of enhanced MSS versus an educational webpage. Aim three (Months 16-60) will assess implementation outcomes and identify contextual factors to facilitate scale-up for future dissemination and implementation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary pathologic stage 0-III cutaneous malignant melanoma
* Three months to five years post-surgery
* No current evidence of cancer
* Not adherent to thorough SSE (i.e., did not check entire body at least once during the past three months)
* ≥ 18 years old
* Internet access
* Able to speak/read English
* Able to provide informed consent

Exclusion Criteria:

* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Body parts examined | Baseline
  Yes/No for a list of body parts examined during most recent SSE in the last three months. This is the primary outcome because SSE thoroughness is associated with detection of thinner tumors. This will be assessed by Reach, Effectiveness, Adoption, Implementation, and Maintenance(RE-AIM) and Practical, Robust Implementation and Sustainability Model (PRISM).
Body parts examined | 3 months
  Yes/No for a list of body parts examined during most recent SSE in the last three months. This is the primary outcome because SSE thoroughness is associated with detection of thinner tumors. This will be assessed by Reach, Effectiveness, Adoption, Implementation, and Maintenance(RE-AIM) and Practical, Robust Implementation and Sustainability Model (PRISM).
Body parts examined | 6 months
  Yes/No for a list of body parts examined during most recent SSE in the last three months. This is the primary outcome because SSE thoroughness is associated with detection of thinner tumors. This will be assessed by Reach, Effectiveness, Adoption, Implementation, and Maintenance(RE-AIM) and Practical, Robust Implementation and Sustainability Model (PRISM).
Body parts examined | 12 months
  Yes/No for a list of body parts examined during most recent SSE in the last three months. This is the primary outcome because SSE thoroughness is associated with detection of thinner tumors. This will be assessed by Reach, Effectiveness, Adoption, Implementation, and Maintenance(RE-AIM) and Practical, Robust Implementation and Sustainability Model (PRISM).
Body parts examined | 18 months
  Yes/No for a list of body parts examined during most recent SSE in the last three months. This is the primary outcome because SSE thoroughness is associated with detection of thinner tumors. This will be assessed by Reach, Effectiveness, Adoption, Implementation, and Maintenance(RE-AIM) and Practical, Robust Implementation and Sustainability Model (PRISM).

SECONDARY OUTCOMES:
Melanoma Diagnosis | 6 months
  This will be assessed by asking the participant at the second follow-up if a melanoma was diagnosed and confirmed by provider via medical records.
Melanoma Diagnosis | 12 months
  This will be assessed by asking the participant at the third follow-up if a melanoma was diagnosed and confirmed by provider via medical records.
Melanoma Diagnosis | 18 months
  This will be assessed by asking the participant at the fourth follow-up if a melanoma was diagnosed and confirmed by provider via medical records.
Melanoma Stage | 3 months
  This will be assessed by asking the participant at the first follow-up what stage melanoma was diagnosed, if diagnosed. Response will be confirmed by provider via medical records.
Melanoma Stage | 6 months
  This will be assessed by asking the participant at the second follow-up what stage melanoma was diagnosed, if diagnosed. Response will be confirmed by provider via medical records.
Melanoma Stage | 12 months
  This will be assessed by asking the participant at the third follow-up what stage melanoma was diagnosed, if diagnosed. Response will be confirmed by provider via medical records.
Melanoma Stage | 18 months
  This will be assessed by asking the participant at the fourth follow-up what stage melanoma was diagnosed, if diagnosed. Response will be confirmed by provider via medical records.
Melanoma Diagnosis Date | 3 months
  This will be assessed by asking the participant at the first follow-up the date of his/her melanoma diagnosis, if diagnosed. Response will be confirmed by provider via medical records.
Melanoma Diagnosis Date | 6 months
  This will be assessed by asking the participant at the second follow-up the date of his/her melanoma diagnosis, if diagnosed. Response will be confirmed by provider via medical records.
Melanoma Diagnosis Date | 12 months
  This will be assessed by asking the participant at the third follow-up the date of his/her melanoma diagnosis, if diagnosed. Response will be confirmed by provider via medical records.
Melanoma Diagnosis Date | 18 months
  This will be assessed by asking the participant at the fourth follow-up the date of his/her melanoma diagnosis, if diagnosed. Response will be confirmed by provider via medical records.
Melanoma Diagnosis | 3 months
  This will be assessed by asking the participant at the first follow-up if a melanoma was diagnosed and confirmed by provider via medical records.

OTHER OUTCOMES:
Age | Baseline
  This will be assessed by asking the participant his/her age in the baseline survey.
Sex | Baseline
  This will be assessed by asking the participant his/her sex in the baseline survey.
Race/Ethnicity | Baseline
  This will be assessed by asking the participant his/her race and ethnicity in the baseline survey.
Education | Baseline
  This will be assessed by asking the participant his/her education level in the baseline survey.
Marital Status | Baseline
  This will be assessed by asking the participant his/her marital status in the baseline survey.
State Residing In | Baseline
  This will be assessed by asking the participant what state he/she resides in the baseline survey.
Employment | Baseline
  This will be assessed by asking the participant his/her employment status in the baseline survey.
Income | Baseline
  This will be assessed by asking the participant his/her income level in the baseline survey.
Health Insurance | Baseline
  This will be assessed by asking the participant if he/she has health insurance coverage in the baseline survey.
Date of Diagnosis | Baseline
  This will be assessed by asking the participant in the baseline survey the date that he/she was diagnosed with skin cancer.
Stage | Baseline
  This will be assessed by asking the participant in the baseline survey the stage of cancer he/she was diagnosed with.
Treatment Received | Baseline
  This will be assessed by asking the participant in the baseline survey what treatment he/she received.
Indoor UV Tanning | 12 months
  This will be assessed by asking the participant in the baseline survey about his/her indoor UV tanning behaviors. Indoor UV tanning is an important covariate because it can pose as a risk factor for melanoma.
Family History of Melanoma | Baseline
  This will be assessed by asking the participant in the baseline survey about his/her family history of melanoma. Family history is an important covariate because it can pose as a risk factor for melanoma.
Month of Assessment | Baseline
  This will be assessed by asking participant in the baseline survey in what month he/she is completing the survey
Month of Assessment | 3 months
  This will be assessed by asking participant in the first follow-up survey in what month he/she is completing the survey
Month of Assessment | 6 months
  This will be assessed by asking participant in the second follow-up survey in what month he/she is completing the survey
Month of Assessment | 12 months
  This will be assessed by asking participant in the third follow-up survey in what month he/she is completing the survey
Month of Assessment | 18 months
  This will be assessed by asking participant in the fourth follow-up survey in what month he/she is completing the survey
Location of Assessment | Baseline
  This will be assessed by asking participant in the baseline survey in what location he/she is completing the survey
Location of Assessment | 3 months
  This will be assessed by asking participant in the first follow-up survey in what location he/she is completing the survey
Location of Assessment | 6 months
  This will be assessed by asking participant in the second follow-up survey in what location he/she is completing the survey
Location of Assessment | 12 months
  This will be assessed by asking participant in the third follow-up survey in what location he/she is completing the survey
Location of Assessment | 18 months
  This will be assessed by asking participant in the fourth follow-up survey in what location he/she is completing the survey
Average UV Index | Baseline
  Assessing the average UV index at solar noon over the 3 months prior to baseline survey submission. This will be determined by the study staff based on the month and location of assessment information provided by the participant in the baseline survey.
Average UV Index | 3 months
  Assessing the average UV index at solar noon over the 3 months prior to the first follow-up survey submission. This will be determined by the study staff based on the month and location of assessment information provided by the participant in the first follow-up survey.
Average UV Index | 6 months
  Assessing the average UV index at solar noon over the 3 months prior to the second follow-up survey submission. This will be determined by the study staff based on the month and location of assessment information provided by the participant in the second follow-up survey.
Average UV Index | 12 months
  Assessing the average UV index at solar noon over the 3 months prior to the third follow-up survey submission. This will be determined by the study staff based on the month and location of assessment information provided by the participant in the third follow-up survey.
Average UV Index | 18 months
  Assessing the average UV index at solar noon over the 3 months prior to the fourth follow-up survey submission. This will be determined by the study staff based on the month and location of assessment information provided by the participant in the fourth follow-up survey.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Manne, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey; Carolyn Heckman, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT05373823/ICF_000.pdf